CLINICAL TRIAL: NCT06346002
Title: Impact of a Mindfulness-based Intervention on Well-being and Mental Health of Elementary School Children: Results From a Randomized Cluster Trial
Brief Title: Impact of a Mindfulness-based Intervention on Well-being and Mental Health of Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bishop's University (Other)
Responsible Party: Principal Investigator, Catherine Malboeuf-Hurtubise, Associate Professor, Bishop's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2026_e_2017
Record Dates: First submitted 2024-03-24; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Mindfulness-based Intervention; Elementary School Children; Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: Randomized cluster trial with a wait-list control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based condition (Experimental): Classes assigned to this condition received the mindfulness-based intervention. The MBI program implemented comprised ten weekly sessions. Activities were drawn from the Mission Méditation program, a MBI intervention specifically tailored for elementary school children. Activities comprised in this intervention encompassed formal (e.g., body scan, sitting, and breathing meditation) and informal meditations (e.g., mindful eating, listening, and touching, mindful walking), as well as positive psychology exercises (e.g., taking care of oneself, gratitude). The weekly sessions, lasting 45 to 60 minutes each, were delivered in a group format by the teachers themselves, in their classroom.
  Interventions: Behavioral: Mindfulness-based intervention
- Wait-list control (No Intervention): Placed on waitlist and then offered the intervention once the data collection phase was over.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — The MBI program implemented comprised ten weekly sessions. Please refer to the arm/group descriptions for further details.
  Arms: Mindfulness-based condition

SUMMARY:
Background: Prevention programs for children such as mindfulness-based interventions (MBIs) are often implemented in schools to prevent psychological disorders from emerging and contribute to children' mental health.

Aim: This study used a randomized cluster design and assessed the impact of a MBI on well-being and mental health of elementary school children's.

Method: 13 elementary school classrooms were randomly allocated to the experimental condition (7 classrooms, n = 127 students) or the waitlist control condition (6 classrooms, n = 104 students). Participants in the experimental condition received a 10-week MBI.

ELIGIBILITY:
Inclusion Criteria:

* Attending the Préville Elementary School
* Spoke sufficient French to fill out questionnaires

Exclusion Criteria:

* Not attending the Préville Elementary School
* Level of French was not good enough to fill out questionnaires

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — All genders were included.
Enrollment: 231 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Symptoms of Mental Health Disorders | Baseline, post-intervention (10 weeks)
  Children completed selected items from the self-report version of the anxiety (three items, e.g., "I worry about little things"), depression (five items, e.g., "Nothing ever goes right for me") and inattention (4 items, e.g., " I forget to do things") subscales of the Behavior Assessment Scale for Children (BASC II)
Basic Psychological Needs Satisfaction | Baseline, post-intervention (10 weeks)
  Participants rated how competent, autonomous, and related they felt in school, by answering a nine-item scale adapted from a scale used in a previous, similar study [57]. Children were asked to rate their agreement with items such as "In school, I feel free to be myself" (autonomy); "I am able to reach my goals" (competence) and "In my relationship with others, I feel appreciated" (relatedness) on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always).
Process Measure | Baseline, post-intervention (10 weeks)
  Finally, participants completed the Mindful Attention and Awareness Scale for Children (e.g., "I find it hard to stay focused on what's happening in the present moment."; [58]) to evaluate pre-to-post changes in their mindfulness abilities. They rated their agreement with each item on a 6-point Likert scale ranging from 1 (never) to 6 (almost always). A higher score on this scale indicates lower levels of mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- École primaire Préville, Saint-Lambert, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request with the PI.